CLINICAL TRIAL: NCT03726931
Title: FES (16α-[18F]-Fluoro-17β-estradiol)-PET: Towards a New Standard to Stage Locally Advanced and Recurrent, Estrogen Receptor Positive (ER+) Breast Cancer? Pilot Study to Compare [18F]FES-PET and [18F]FDG-PET
Acronym: FORESIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, C. Menke- van der Houven van Oordt, MD PhD, Medical Oncologist and Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018.451
Record Dates: First submitted 2018-10-16; First posted 2018-11-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: In this multicenter observational study with invasive measurements, patients with clinically ER+/HER2- LABC and LRR breast cancer will be included. All patients will undergo the current 'standard' diagnostic procedures including a histological biopsy of the primary tumor, cytology of axillary lymph nodes and imaging procedures with mammography, ultrasound of breast and axilla, magnetic resonance imaging (MRI) breast and whole body [18F]FDG PET combined with diagnostic chest/abdominal CT. In addition, all patients will undergo the 'experimental' imaging procedure with [18F]FES PET/CT. After evaluation of the obtained scans (independently for both scans), an 'experimental histological biopsy' of a lymph node metastasis will be obtained and clinically relevant [18F]FDG+ and/or [18F]FES+ lesions and/or suspicious lesions on CT will be biopsied according to standard clinical practice for pathological analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [18F]FES (Experimental): All patients will receive an additional PET/CT scan: [18F]FES PET/CT scan.
  Interventions: Diagnostic Test: 18F-Fluorestradiol PET/CT scan

INTERVENTIONS:
Diagnostic Test: 18F-Fluorestradiol PET/CT scan — [18F]FES PET/CT scan will be performed after administration of radioactive labelled estrogen.
  Other Names: [18F]FES PET/CT scan

SUMMARY:
Accurate staging is of great importance in patients with clinically locally advanced primary breast cancer (LABC, stage III) or locoregional recurrent (LRR) breast cancer for making a correct treatment plan. According to current guidelines, staging is performed with positron emission tomography (PET) using the 2-[18F]fluoro-2-deoxy-D-glucose ([18F]FDG) PET tracer, combined with diagnostic computed tomography (CT). However, previous studies have shown that this technique (with the current PET tracer) might not be sufficient for accurate staging. Specifically in low grade, estrogen receptor positive (ER+) breast cancer metastases can be missed due to the low metabolic activity, leading to low uptake of [18F]FDG. Therefore, there is a clinical need to improve staging procedures. 16α-[18F]-fluoro-17β-estradiol ([18F]FES), an ER-targeted PET tracer, allows imaging of ER+ tumor lesions regardless of their metabolic activity. Patients with clinically LABC and LRR have a 25-50% risk of distant metastases. Correct identification of distant metastases allows adaptation of the treatment plan to avoid burdensome treatment with surgery, systemic and radiotherapy in order to maintain quality of life. In case of oligometastases, correct identification increases the likelihood for cure with local treatment. In the current study we will compare disease staging with [18F]FES- and [18F]FDG PET in patients with clinically LABC/LRR breast cancer. Objective: To determine whether [18F]FES PET/CT improves staging for women with clinically LABC or LRR, ER+/HER2- breast cancer as compared to standard [18F]FDG PET/CT. Study design: Multicenter prospective study with invasive measurements. Study population: 20 LABC and 20 LRR ER+/HER2- breast cancer patients. Main study parameters/endpoints: To determine the percentage of patients with a correctly changed treatment plan according to information obtained from [18F]FES PET/CT compared to [18F]FDG PET/CT at staging and at 6 months of follow-up; to determine the percentage of metastatic lesions detected and missed with [18F]FES PET/CT compared to [18F]FDG PET/CT (at staging and during follow-up). Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will receive an intravenous cannula for tracer injection and blood sampling, causing potentially transient discomfort at the site of the cannula insertion. Tumor biopsy will be performed from an easy accessible lesion and the most frequent complications that can occur are discomfort, bleeding and (local) infection. The risk of complications from a tumor biopsy is considered low: 0.24-1.6% and 0.11-0.48% for major complications and mortality, respectively. Radiation exposure from a [18F]FES PET and [18F]FDG PET scan usually ranges between 4-11 mSv and 7-8 mSv, respectively. Radiation exposure from a diagnostic CT scan ranges between 8-14 mSv. The total radiation burden is considered justifiable when compared to the information that can be obtained from this study, in this patient group with breast cancer. Imaging with [18F]FES PET may improve staging for patients with breast cancer as it may show tumor lesions that could not be identified with [18F]FDG PET, the current standard for staging. If this is the case, the initial treatment goal and intensity can be adjusted which can have beneficial effects for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Clinically LABC (stage III) or LRR breast cancer (all histological types) with ER+, HER2- and low grade according to Bloom Richardson criteria (grade 1-2)
* Females aged 18 years or older at screening
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-2
* Candidates for treatment with curative intent (patients are also allowed for inclusion in the current study if they have undergone recent surgery (<6 weeks) for current breast cancer and require staging because of unexpected stage III disease)
* In case [18F]FDG PET/CT has already been performed, patients can be included <21 days after this scan
* Estimated glomerular filtration rate (eGFR) ≥30 ml/min
* Written and signed informed consent

Exclusion Criteria:

* History with another cancer within the last 5 years, except non-melanoma skin cancer
* Undergoing treatment for current breast cancer such as (neo)adjuvant chemotherapy, hormonal therapy (only in case of Tamoxifen), radiotherapy or investigational drug therapy
* Pregnancy or lactating women
* Any medical, psychological or social condition that may interfere with the subject's safety and participation in the study, will lead to exclusion from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2023-01-29 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a correctly changed treatment plan according to [18F]FES PET/CT compared to [18F]FDG PET/CT. | 2 years
  Percentage of patients with a correctly changed treatment plan according to information obtained with [18F]FES PET/CT compared to [18F]FDG PET/CT at staging.
Percentage of metastatic lesions detected with [18F]FES PET/CT compared to [18F]FDG PET/CT. | 2 years
  Percentage of metastatic lesions detected with [18F]FES PET/CT compared to [18F]FDG PET/CT at staging.
Percentage of missed metastases with [18F]FES PET/CT compared to [18F]FDG PET/CT. | 2 years
  Percentage of missed metastases with [18F]FES PET/CT compared to [18F]FDG PET/CT (at staging and developed during follow-up).
Percentage of correct treatment plans as well as diagnostic confidence after 6 months of follow-up based on the added information obtained with [18F]FES PET/CT compared to [18F]FDG PET/CT. | 2 years
  Percentage of correct treatment plans as well as diagnostic confidence after 6 months of follow-up as determined by the adjudication committee based on the added information obtained with [18F]FES PET/CT compared to [18F]FDG PET/CT.

SECONDARY OUTCOMES:
[18F]FES/[18F]FDG uptake related to size of the lesion | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to size of the lesion.
[18F]FES/[18F]FDG uptake related to location of the lesion. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to location of the lesion.
[18F]FES/[18F]FDG uptake related to histological subtype. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to histological subtype.
[18F]FES/[18F]FDG uptake related to grade. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to grade.
[18F]FES/[18F]FDG uptake related to ER expression level. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to ER expression level.
[18F]FES/[18F]FDG uptake related to PR expression level. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to PR expression level.
[18F]FES/[18F]FDG uptake related to HER2 expression level. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to HER2 expression level.
[18F]FES/[18F]FDG uptake related to Ki67%/mitotic index. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to Ki67%/mitotic index.
[18F]FES/[18F]FDG uptake related to intensity of ER staining. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to intensity of ER staining.
[18F]FES/[18F]FDG uptake related to intensity of tumor cell density. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to intensity of tumor cell density.
[18F]FES/[18F]FDG uptake related to intensity of microvessel density. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to intensity of microvessel density.
[18F]FES/[18F]FDG uptake related to infiltration of lymphocytes. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to infiltration of lymphocytes.
[18F]FES/[18F]FDG uptake related to amount of necrosis. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to amount of necrosis.
[18F]FES/[18F]FDG uptake related to amount of stroma. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to amount of stroma.
[18F]FES/[18F]FDG uptake related to expression of glucose transporter-1 (GLUT1) in the primary tumor, lymph node and distant metastases. | 2 years
  [18F]FES/[18F]FDG uptake in the primary tumor, lymph node and distant metastases will be related to expression of glucose transporter-1 (GLUT1) in the primary tumor, lymph node and distant metastases.
Cut off value for [18F]FDG SUV max below which [18F]FES PET/CT adds information for staging. | 2 years
  Cut off value for [18F]FDG SUV max below which [18F]FES PET/CT adds information for staging.
Cut off value for [18F]FDG SUV peak below which [18F]FES PET/CT adds information for staging. | 2 years
  Cut off value for [18F]FDG SUV peak below which [18F]FES PET/CT adds information for staging.
Cut off value for grade below which or above which [18F]FES PET/CT adds information for staging. | 2 years
  Cut off value for grade below which or above which, respectively, [18F]FES PET/CT adds information for staging.
Cut off value for ER expression level below which or above which [18F]FES PET/CT adds information for staging. | 2 years
  Cut off value for ER expression level below which or above which [18F]FES PET/CT adds information for staging.

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iqbal R, Menke-van der Houven van Oordt CW, Oprea-Lager DE, Booij J. [18F]FES uptake in the pituitary gland and white matter of the brain. Eur J Nucl Med Mol Imaging. 2021 Aug;48(9):3009-3010. doi: 10.1007/s00259-021-05281-8. Epub 2021 Mar 17. No abstract available. PMID 33730173